CLINICAL TRIAL: NCT01448265
Title: Real-Time Assessment of Cryoballoon Pulmonary Vein Isolation Using a Novel Circular Mapping Catheter
Acronym: CRYO-MAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dierk Thomas, M.D., Assistant Professor, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRYO-MAP
Record Dates: First submitted 2011-09-30; First posted 2011-10-07 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; circular mapping catheter; cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paroxysmal atrial fibrillation. (Experimental)
  Interventions: Procedure: Cryoballoon ablation.

INTERVENTIONS:
Procedure: Cryoballoon ablation. — Cryoballoon ablation using a novel circular mapping catheter.

SUMMARY:
Background: Atrial fibrillation (AF) is the most frequent sustained cardiac arrhythmia, impairs quality of life and increases stroke risk and mortality. Recent clinical experience with the Arctic Front™ cryoballoon ablation catheter system (Medtronic) suggests that it can be used to isolate the pulmonary veins (PVs) safely and effectively in patients with AF, thereby eliminating the recurrence of AF.

Hypothesis: Our hypotheses are (1) that visualization of real-time pulmonary vein conduction during cryoballoon ablation of atrial fibrillation using a novel spiral circumferential mapping catheter (Achieve™) is feasible and safe, and (2) that procedure and fluoroscopy times decrease with experience.

Objective: The purpose of this study is to assess safety, feasibility, and a learning curve associated with cryoballoon catheter ablation using a novel circular mapping catheter (Achieve™, Medtronic) inserted through the lumen of the cryoballoon in patients with symptomatic paroxysmal atrial fibrillation.

The primary goal is to evaluate successful pulmonary vein isolation using the Achieve™ mapping catheter. The reduction of procedure and fluoroscopy times during the first 40 patients treated with this approach will be analyzed to evaluate a potential learning curve upon introduction of the technique.

DETAILED DESCRIPTION:
A total of 40 patients scheduled for a first ablation of paroxysmal AF will be included. All study subjects will undergo cryoablation using the 28 mm Arctic Front™ Cryoablation Catheter. A double transseptal approach will be followed in all study patients, allowing for use of regular guide wire and circular mapping catheter, respectively, if required.

Use of the 20 mm Achieve™ circular mapping catheter is preferred. The 15 mm AchieveTM catheter may be used at the physician's discretion. If stable balloon positions cannot be obtained, the Achieve™ catheter will be replaced by a regular guide wire and pulmonary vein isolation will be assessed by a circular mapping catheter (Lasso™; Biosense Webster) introduced through a second transseptal puncture. Cryoablations will be applied for 5 minutes each. Premature terminations will be allowed at the physician's discretion but should be avoided to allow for detection of late pulmonary vein isolation during cryoenergy application. Cryoballoon catheter manipulations (e.g., pull down maneuver) may be performed during energy application. During ablation of septal pulmonary veins, electrical phrenic nerve stimulation will be performed to exclude phrenic nerve palsy. If additional single point ablations are required to achieve electrical isolation of pulmonary veins, a linear cryocatheter (Freezor™ Max; Medtronic) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal atrial fibrillation
* ≥18 and ≤75 years of age
* Failure of one or more antiarrhythmic drugs
* Referral for a pulmonary vein isolation catheter ablation procedure to treat atrial fibrillation

Exclusion Criteria:

* Previous ablation of atrial fibrillation
* Documented left atrial thrombus
* Irregular pulmonary vein anatomy according to transesophageal echocardiography
* Atrial fibrillation secondary to reversible cause
* Amiodarone therapy in the previous 6 months
* Cardiac surgery within the prior 6 months
* Myocardial infarction within the previous 2 months
* Ejection fraction < 40%
* NYHA class III or IV
* Moderate to severe valvular heart disease
* Previous valve replacement
* Pacemaker or implantable cardioverter defibrillator placement in the prior 3 months
* History of stroke or TIA within the previous 12 months
* Left atrial size ≥ 50 mm
* Contraindication for anticoagulation medication
* Life expectancy of less than 12 months
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Feasibility, defined as successful pulmonary vein isolation using the novel circular mapping catheter with the cryoballoon. | Participants will be followed for the duration of the ablation procedure, an expected average of 1-3 hours.

SECONDARY OUTCOMES:
Time from beginning of the freeze to conduction blockade ("time to effect"). | Participants will be followed for the duration of the ablation procedure, an expected average of 1-3 hours.
Treatment-related adverse events. | Participants will be followed for the duration of the ablation procedure, an expected average of 1-3 hours.
Procedure time. | Participants will be followed for the duration of the ablation procedure, an expected average of 1-3 hours.
Overall fluoroscopy time and dose. | Participants will be followed for the duration of the ablation procedure, an expected average of 1-3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Thomas, MD, Principal Investigator — Department of Cardiology, University of Heidelberg
Locations (1):
- Department of Cardiology, University of Heidelberg, Heidelberg, Germany